CLINICAL TRIAL: NCT03536598
Title: A Double-blind, Randomized, Multi-center Phase III Clinical Trial to Evaluate the Safety and Efficacy of CJ-30060 Compared With Amlodipine/Valsartan Combination Therapy and Valsartan/Rosuvastatin Combination Therapy in Hypertensive Patients With Hyperlipidemia
Brief Title: Study to Evaluate the Safety and Efficacy of CJ-30060 in Hypertensive Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_EXR_301
Record Dates: First submitted 2017-07-18; First posted 2018-05-24 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2017-07

CONDITIONS: Hypertension With Hyperlipidemia
MeSH Terms: interventions — Amlodipine; Valsartan; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): Amlodipine 10mg + Valsartan 160mg + Rosuvastatin 20mg
  Interventions: Drug: Amlodipine 10 mg + Valsartan 160 mg + Rosuvastatin 20 mg
- Reference 1 (Active Comparator): Amlodipine 10mg + Valsartan 160mg
  Interventions: Drug: Amlodipine 10 mg + Valsartan 160 mg
- Reference 2 (Active Comparator): Valsartan 160mg + Rosuvastatin 20mg
  Interventions: Drug: Valsartan 160 mg + Rosuvastatin 20 mg

INTERVENTIONS:
Drug: Amlodipine 10 mg + Valsartan 160 mg + Rosuvastatin 20 mg
  Arms: Test
Drug: Amlodipine 10 mg + Valsartan 160 mg
  Arms: Reference 1
Drug: Valsartan 160 mg + Rosuvastatin 20 mg
  Arms: Reference 2

SUMMARY:
To evaluate the safety and efficacy of CJ-30060 compared with amlodipine/valsartan combination therapy and valsartan/rosuvastatin combination therapy in hypertensive patients with hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 74 years
* Patient with dyslipidemia and hypertension

Exclusion Criteria:

* At screening, siSBP ≥ 200 mmHg or siDBP ≥ 120mmHg or LDL-C > 250mg/dL or TG ≥ 400mg/dL
* At screening, siSBP difference is ≥ 20 mmHg or siDBP difference is ≥10 mmHg
* Secodary hypertension
* Type I or uncontrolled diabetes mellitus (HbA1c ≥ 9 %)

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Change of LDL-C and siSBP | baseline and 8 weeks
  Mean change from baseline in LDL-C and siSBP at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ju Choi, Ph.D, Principal Investigator — Seoul National University Bundang Hospital